CLINICAL TRIAL: NCT00827437
Title: Family-Staff Communication Intervention at the Time of Difficult Treatment Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Pamela S. Hinds PhD, RN, St. Jude Children's Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DECID4
Record Dates: First submitted 2008-08-06; First posted 2009-01-22 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2011-06

CONDITIONS: Difficult Decision Making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Other: Parent Interview

INTERVENTIONS:
Other: Parent Interview — To include the PI, Nursing Research Specialist,Clinical Research Associate or Clinical Nurse Specialist

SUMMARY:
The primary aim of this single site study was to assess the feasibility of implementing a staff/parent communication intervention within 72 hours of the parents making an end-of-life decision on behalf of their child.

DETAILED DESCRIPTION:
Parents/guardians of children with incurable cancer face end-of-life decisions on behalf of their child including whether or not to enroll their child in a Phase I study, whether or not to agree to a 'do not resuscitate' status, or to begin terminal care. Descriptive research to date indicates that one of the factors that most helps parents to make these decisions and to remain satisfied with the decision afterward is their perception that they decided as a 'good parent' would decide. Parents define being a 'good parent' as making a decision that is in the best interest of their child. Parents' perception of their success in being a good parent is influenced by their interactions with the child's health care providers. Health care providers who are not fully informed about the decision and the parents' rationale for the decision are likely to convey doubt about the decision to parents and to other health care providers. Parents interpret this doubt as staff questioning the parents' ability to make good decisions. Lack of adequate information also creates staff tension. This single-site feasibility study will implement and evaluate a two-part communication intervention designed to identify parents' definition of being a good parent, and to communicate this definition and the rationale for the parents' decision to staff. The intervention will be implemented in 60 to 80 end-of-life clinical care situations in which parents have made a decision on behalf of a child who is still living. The feasibility study is guided by the Pediatric Quality of Life at End of Life model. The parent/guardian intervention includes a face-to-face interview with parents regarding their definition of a 'good parent' and their basis for the decision they made. Parents/guardians will be interviewed within 72 hours after making the end of life decision and again 1 to 3 weeks after making the decision. Health care professionals assigned to the terminally ill child will receive the communication intervention within hours of the parent interview, and will evaluate its usefulness 1 to 2 weeks after receiving it.

1.1 To assess the feasibility of delivering the two-part communication intervention. The definition of feasible is that 50% of all interventions are successfully implemented.

1.1.1 To identify all three types of difficult treatment decisions within the defined time frame (thus identifying eligible parents/guardians and obtaining consent within 72 hours after the decision was made), document the study team's ability to successfully implement the intervention before the child's death (obtaining the parent/guardian information and sharing that with the defined staff such that the family achieves the definition of being fully evaluable as a study participant), and document the participation rate by tracking the number of eligible parents/guardians who agree to participate, decline to participate or withdraw from the study.

1.2: To assess staff perceptions of the impact of the communication intervention on staff 1 to 2 weeks after the intervention.

1.2.1 to measure: a) staff recall of the definition of a good parent and the rationale for the decision; b) staff perception of how this knowledge influenced their care for the family; c) staff satisfaction with the verbal and written communication intervention forms; and d) the impact of the communication intervention on team tension and team communication about the parents' decisions.

1.3: To assess the impact of the communication on parents/guardians by recording their perceptions of the positive and negative aspects of the intervention at the time of the intervention and 1 to 3 weeks after the decision making.

ELIGIBILITY:
Inclusion Criteria:

* Eligible parents/guardian can be enrolled only one time and will be:
* 21 years of age and older.
* This study will enroll only parents/guardians who are 21 years of age and older. The investigators clinical experience is that when the parent/guardian is younger, additional adult members of the family are involved in the decision making and that asking a single person to identify him or herself as the primary parent/guardian creates difficulties for the family.
* As a result, no parent/guardian younger than age 21 will be enrolled in this study.
* English-speaking.
* Willing to give written consent to participate.
* The parents/guardians of a child with incurable cancer or a fatal cancer-related condition who is being treated at St. Jude Children's Research Hospital
* The parents/guardians who made an end-of-life decision on behalf of the seriously ill child within the previous 72-hours.
* Eligible staff can be enrolled more than one time and will be:
* English-speaking
* Willing to give written consent to participate

Exclusion Criteria:

* Parents/guardians who meet the above criteria but are identified by their attending or social support staff member (an assigned social worker or psychologist at St. Jude Children's Research Hospital) as emotionally or mentally unable to participate in the informed consent process will not be approached about participating in the study.
* Parents who are identified by their attending or social support staff member as likely to find the study too burdensome because of their emotional or mental state.
* Parents who did not make the end-of-life decision (i.e., when the patient made the decision).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2004-01; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of delivering the two-part communication intervention. The definition of feasible is that 50% of all interventions are successfully implemented. | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Hinds, PhD, RN, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org